CLINICAL TRIAL: NCT05005494
Title: Study of the Hypnotic and Anti-nociceptive Components of Magnesium Using Electroencephalogram Spectral Entropy and Pupillometry During Total Intravenous General Anaesthesia
Brief Title: Hypnotic and Anti-nociceptive Components of Magnesium
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Head of Anesthesiology Departement, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MG-Entropy
Record Dates: First submitted 2021-07-27; First posted 2021-08-13 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: Double blinded prospective randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient, anesthesiologist and surgeon are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium sulfate IV (Active Comparator): 10 patients scheduled for thyroidectomy
  Interventions: Drug: Magnesium sulfate IV
- Placebo (Placebo Comparator): 10 patients scheduled for thyroidectomy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium sulfate IV — Infusion of magnesium sulphate 50 mg/kg (eq. 0.5ml/kg of magnesium sulphate 100mg/ml)
  Arms: Magnesium sulfate IV
Drug: Placebo — Infusion of NaCl (sodium chloride) 0.9% (placebo eq. 0.5ml/kg of NaCl 0.9%)
  Arms: Placebo

SUMMARY:
The aim of our study is to evaluate the effect of magnesium on the hypnotic effect of propofol.

DETAILED DESCRIPTION:
The aim of our study is to evaluate the effect of magnesium on the hypnotic effect of propofol. To achieve this, the investigators will analyse the effect of magnesium on the brain concentrations of propofol required to achieve a State Entropy value between 50-60, which corresponds to the recommended depth of anaesthesia. Our study will also evaluate the intraoperative anti- nociceptive effect of magnesium using pupillometry and its two indices, PPI and PRD

ELIGIBILITY:
Inclusion Criteria:

* Adult > 18 years
* Patients of both sexes
* Any patient scheduled for thyroidectomy at the University Hospital of Liege

Exclusion Criteria:

* Heart failure with left ventricular ejection fraction < 35
* Renal insufficiency (clearance < 40 mL/min)
* Neuromuscular diseases
* Atrioventricular block
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Propofol target concentration | through study completion, an average of 3 months
  The target concentration of Propofol TCI (target-control infusion) to achieve a state entropy value between 50-60

SECONDARY OUTCOMES:
Morphine consumption | through study completion, an average of 3 months
  Morphine consumption titrated in the recovery room and morphine equivalents claimed during the first 24 hours postoperatively
PPI Measure | through study completion, an average of 3 months
  PPI (pupillary pain index) by pupillometry with "AlgiScan®" monitoring, before endotracheal intubation and with a State Entropy of 50-60, then every 5 min between endotracheal intubation and surgical incision
PRD Measure | through study completion, an average of 3 months
  PRD (pupillary reflex dilatation) during laryngoscopy maintained for 30 sec, surgical incision and 10min after surgical incision

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Liege,, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No